CLINICAL TRIAL: NCT05022446
Title: The Impact of COVID-19 on Pulmonary Procedures: A Nationwide Survey
Brief Title: The Impact of COVID-19 on Pulmonary Procedures
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0662; NCI-2021-01788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0662 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-18; First posted 2021-08-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete survey over 5-10 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates the changes in practice by pulmonary procedural programs across the United States as they faced the coronavirus pandemic. Information gathered from this study may help guide pulmonary programs on a wider scale and improve their practice. The study may also help researchers understand where they should focus research efforts to better respond to a pandemic in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess how pulmonary medicine programs adapted their procedural practices and techniques, ambulatory operations, and provider staffing in response to the coronavirus-2019 (COVID-19) epidemic.

OUTLINE:

Participants complete survey over 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonologists that are members of the American Association of Bronchology and Interventional Pulmonology (AABIP) and/or the American College of Chest Physicians (ACCP)
* These organizations were chosen because their member databases are composed of pulmonologists in the United States (U.S.) that perform the pulmonary procedures described in this survey. Letters of approval will be obtained from these organizations and provided to the MD Anderson Institutional Review Board (IRB). Once the MD Anderson IRB approves this survey study, the survey will be sent to the relevant subcommittees of these organizations for their electronic dissemination to their membership

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonologists that are members of the American Association of Bronchology and Interventional Pulmonology (AABIP) and/or the American College of Chest Physicians (ACCP)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the pulmonary medicine programs adapted that their procedural practices in response to the coronavirus-2019 (COVID-19) epidemic. | through study completion, an average of 1 year
To evaluate the pulmonary medicine programs that adapted their provider staffing in response to the coronavirus-2019 (COVID-19) epidemic. | through study completion, an average of 1 year
To evaluate the pulmonary medicine programs that adapted their techniques in response to the coronavirus-2019 (COVID-19) epidemic. | through study completion, an average of 1 year
To evaluate the pulmonary medicine programs that adapted their ambulatory operations in response to the coronavirus-2019 (COVID-19) epidemic. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruce F Sabath, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org